CLINICAL TRIAL: NCT07274696
Title: A Multicenter, Open-Label, Randomized, Placebo-Controlled Study Protocol on the Effect of Mecobalamin in Promoting Recurrent Laryngeal Nerve Function Recovery After Thyroid Surgery（MIREN Trial）
Brief Title: Mecobalamin in Promoting Recurrent Laryngeal Nerve Function Recovery After Thyroid Surgery
Acronym: MIREN
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: West China Tianfu Hospital, Sichuan University (Unknown); Shang Jin Hospital of West China Hospital,Sichuan University (Unknown); Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, China (Unknown); Sanya People's Hospital (Unknown)
Responsible Party: Principal Investigator, Yu Feng, West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025(2153)
Record Dates: First submitted 2025-11-25; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Patients Undergoing Open Thyroid Surgery
Keywords: thyroid surgery; recurrent laryngeal nerve; mecobalamin
MeSH Terms: interventions — mecobalamin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mecobalamin Group (Experimental): The patient began taking mecobalamin tablets orally within 24 hours after thyroid surgery, three times a day, 0.5mg each time, for three consecutive months.
  Interventions: Drug: Mecobalamin
- Control group (Placebo Comparator): The patient was given a placebo within 24 hours after thyroid surgery, which was identical in appearance, size, color, dosage form, weight, taste, and smell to mecobalamin tablets, three times a day, 0.5mg each time, for three consecutive months.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mecobalamin — The patient began taking mecobalamin tablets orally within 24 hours after thyroid surgery, three times a day, 0.5mg each time, for three consecutive months.
  Arms: Mecobalamin Group
Drug: placebo — The patient was given a placebo within 24 hours after thyroid surgery, which was identical in appearance, size, color, dosage form, weight, taste, and smell to mecobalamin tablets, three times a day, 0.5mg each time, for three consecutive months.
  Arms: Control group

SUMMARY:
Recurrent laryngeal nerve injury is one of the most common and serious complications affecting quality of life after thyroid surgery. Intraoperative traction, clamping, thermal injury, or direct transection can lead to its dysfunction. Unilateral injury causes vocal cord paralysis, manifesting as hoarseness, coughing while drinking, and vocal fatigue; bilateral injury can result in severe dyspnea, potentially requiring tracheotomy and posing life-threatening risks. Although intraoperative neuromonitoring has reduced the risk of permanent injury, temporary nerve palsy remains very common, imposing a dual physiological and psychological burden on patients. Therefore, exploring safe and effective methods to promote the recovery of recurrent laryngeal nerve function postoperatively is an urgent clinical issue in thyroid surgery.

As a motor nerve, the functional recovery of the recurrent laryngeal nerve depends on axonal regeneration and reinnervation of the laryngeal muscles. This process is slow and often incomplete, influenced by factors such as the extent of injury and patient age. Current clinical management of postoperative recurrent laryngeal nerve palsy primarily involves conservative observation and voice training, lacking proactive pharmacological interventions. This presents a clear rationale and clinical entry point for research.

Mecobalamin, the active form of vitamin B12, has high bioavailability and directly participates in methylation reactions, as well as nucleic acid and protein synthesis. Studies have confirmed its multifaceted role in treating peripheral neuropathy: (1) It promotes myelin regeneration by enhancing Erk1/2 and Akt activity, accelerating the myelination of damaged nerve fibers; (2) It enhances nerve regeneration by promoting the synthesis and secretion of nerve growth factors; (3) It improves nerve cell metabolism and repairs damaged nerve cell membranes; (4) It exerts neurotrophic effects by stimulating the proliferation and activity of Schwann cells, thereby increasing the secretion of neurotrophic factors and optimizing the microenvironment for nerve regeneration.

Although mecobalamin is theoretically beneficial for nerve repair and has been successfully applied in other neuropathies, high-quality clinical studies specifically targeting its use for recurrent laryngeal nerve recovery after thyroid surgery are still lacking. Existing literature consists mostly of small-sample retrospective analyses or case reports with inconsistent conclusions and limitations such as selection bias and inadequate control of confounding factors. There is a lack of large-sample, multicenter, randomized controlled trials to provide high-level evidence-based medical data.

Based on this background, the investigators plan to conduct a nationwide multicenter, randomized controlled study. The primary endpoint will be objective acoustic parameters measured by computerized voice analysis, while secondary endpoints will include patient-reported quality of life outcomes, time to voice recovery, subjective patient satisfaction, incidence of permanent paralysis, and adverse drug reactions. The study aims to scientifically and objectively evaluate the efficacy and safety of mecobalamin in promoting the recovery of recurrent laryngeal nerve function after thyroid cancer surgery, providing new therapeutic strategies to optimize perioperative management and improve the quality of life for patients.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, randomized controlled trial. Inclusion Criteria: (1) Patients aged 18-75 years (inclusive); (2) Scheduled to undergo thyroid surgery (including thyroid gland and isthmus resection, total thyroidectomy, etc.); (3) Preoperative laryngoscopy confirms normal bilateral vocal cord mobility; (4) Intraoperative neuromonitoring (IONM) technology is used in all cases; (5) Voluntarily and capable of providing signed informed consent. Exclusion Criteria: (1) Pre-existing hoarseness or recurrent laryngeal nerve palsy; (2) Planned surgery limited to the thyroid isthmus only, or the isthmus plus the medial one-third of both lobes; (3) Pre-existing severe peripheral neuropathy due to other causes (e.g., diabetes mellitus, alcoholism); (4) Pregnant or lactating women; (5) Chronic use of high-dose vitamin B12 or other neurotrophic drugs; (6) Conditions interfering with drug administration or absorption (e.g., dysphagia, intestinal obstruction); (7) Severe pre-existing comorbidities with intolerance to general anesthesia or surgery; (8) History of vitamin B12 allergy; (9) Concurrent participation in another clinical study that may interfere with this trial.

Eligible patients will be randomly assigned in a 1:1 ratio to either the experimental group (Mecobalamin group) or the control group (control group). Data to be collected includes: (1) Basic Information: Name, randomization number, treating hospital, hospital admission number, group assignment, phone number, age, height, weight, BMI, comorbidities (cardiovascular, endocrine, thyroid diseases, etc.); (2) Preoperative Imaging and Laboratory Data: Laryngoscopy results, thyroid ultrasound, electrocardiogram (ECG), TSH, FT3, FT4, TT3, TT4, Tg, TgAb; (3) Surgical Data: Diagnosis, operating surgeon, surgical procedure, surgery date, intraoperative complications, intraoperative signal changes of the vagus nerve, recurrent laryngeal nerve, and superior laryngeal nerve; (4) Voice Assessments (Preoperative, Postoperative Day 1, Postoperative 1 month, 3 months, 6 months): Objective acoustic parameters of voice quality, Voice Handicap Index-10 (VHI-10), Voice-Related Quality of Life-10 (V-RQOL-10), subjective perceptual evaluation of voice quality (GRBAS scale); (5) Postoperative Pathological Results: Postoperative pathological TNM staging, postoperative pathological diagnosis, postoperative treatment; (6) Surgical Complications: Whether secondary surgery was required due to complications; (7) Postoperative Mecobalamin/Placebo Usage: Dosage, course duration, adverse drug events.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-75 years (inclusive) Scheduled to undergo thyroid surgery (including thyroid gland and isthmus resection, total thyroidectomy, etc.) Preoperative laryngoscopy confirms normal bilateral vocal cord mobility Intraoperative neuromonitoring (IONM) technology is used in all cases Voluntarily and capable of providing signed informed consent.

Exclusion Criteria:

Pre-existing hoarseness or recurrent laryngeal nerve palsy Planned surgery limited to the thyroid isthmus only, or the isthmus plus the medial one-third of both lobes Pre-existing severe peripheral neuropathy due to other causes (e.g., diabetes mellitus, alcoholism) Pregnant or lactating women Chronic use of high-dose vitamin B12 or other neurotrophic drugs Conditions interfering with drug administration or absorption (e.g., dysphagia, intestinal obstruction) Severe pre-existing comorbidities with intolerance to general anesthesia or surgery History of vitamin B12 allergy Concurrent participation in another clinical study that may interfere with this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Jitter | Preoperative, within two weeks after surgery, 1 month postoperative, 3 months postoperative, and 6 months postoperative
  Jitter reflects the regularity of the voice in terms of frequency. A smaller jitter value indicates higher regularity of the voice in terms of frequency.
Shimmer | Preoperative, within two weeks after surgery, 1 month postoperative, 3 months postoperative, and 6 months postoperative
  Shimmer reflects the regularity of the voice in terms of amplitude. A smaller shimmer value indicates higher regularity of the voice in terms of amplitude.
Fundamental frequency (F0) | Preoperative, within two weeks after surgery, 1 month postoperative, 3 months postoperative, and 6 months postoperative
Maximum Phonational Frequency Range (MPFR) | Preoperative, within two weeks after surgery, 1 month postoperative, 3 months postoperative, and 6 months postoperative
  The frequency range from the lowest to the highest pitch a person can produce (in Hz or semitones).
Noise-to-Harmonic Ratio (NHR) | Preoperative, within two weeks after surgery, 1 month postoperative, 3 months postoperative, and 6 months postoperative
  The NHR parameter is the ratio of non-harmonic components within the 1,500-4,500 Hz range to harmonic components within the 70-4,500 Hz range. It can be used to assess the proportion of noise components in the voice.

SECONDARY OUTCOMES:
The Voice Handicap Index-10 (VHI-10) | Preoperative, 1 day postoperative, 1 month postoperative, 3 months postoperative, and 6 months postoperative
  The VHI-10 is a voice disorder index scale containing 10 items, comprising 5 functional items, 3 physical items, and 2 emotional items. Each item is scored from 0 to 4, with different scores representing the frequency of occurrence for that item: "Never" is 0 points; "Almost Never" is 1 point; "Sometimes" is 2 points; "Almost Always" is 3 points; and "Always" is 4 points. A higher score indicates a greater impact of the voice disorder in that domain and a more severe self-assessment of the voice disorder by the subject. The critical value for the VHI-10 is 8 points, and subjects with a VHI score ≥ 8 are classified as having a voice disorder.
The Voice-Related Quality of Life (V-RQOL-10) scale | Preoperative, 1 day postoperative, 1 month postoperative, 3 months postoperative, and 6 months postoperative
  Consists of 10 items, encompassing two domains: social-emotional and physical-functioning. The items describe the subjective experiences of patients with voice disorders. Severity is rated on a 5-point scale, where 1 represents "none," 2 represents "a little," 3 represents "a moderate amount," 4 represents "a lot," and 5 represents "a great deal." This questionnaire uses "reverse scoring," and the final scores need to be transformed to a 0 to 100 scale. A higher overall score indicates better voice-related quality of life, while a lower score indicates worse voice-related quality of life.
The subjective auditory-perceptual assessment of voice quality (GRBAS Scale) | Preoperative, 1 day postoperative, 1 month postoperative, 3 months postoperative, and 6 months postoperative
  This scale consists of five parameters: overall grade of hoarseness (G), roughness (R), breathiness (B), asthenia (A), and strain (S). Each parameter is rated on a severity scale from 0 to 3: 0 indicates normal, 1 indicates mild deviation, 2 indicates moderate deviation, and 3 indicates severe deviation. A higher score represents a more severe voice disorder. The assessment is conducted by professional audiologists, voice specialists, and the patient's family members.
Stroboscopy | Preoperative, If necessary after surgery
  This examination utilizes the principle of persistence of vision to observe the vocal cords in a seemingly stationary or slow-motion vibrating state through visual superposition. Dynamic laryngoscopy is performed preoperatively, and the stroboscopic findings are recorded. Postoperatively, it is conducted on patients presenting with voice abnormalities, dysphonia, or suspected abnormal vocal cord mobility to confirm the mobility of the vocal cords.
Intraoperative neural signals | Intraoperative
  During the surgery, IONM technology was used to monitor neural signals from the vagus nerve, recurrent laryngeal nerve, and superior laryngeal nerve both before and after nerve exposure.
The Eating Assessment Tool (EAT-10) | Preoperative, 1 day postoperative, 1 month postoperative, 3 months postoperative, and 6 months postoperative
  This instrument consists of 10 questions, with severity rated on a scale from 0 to 4. A score of 0 indicates "no problem," 1 indicates "mild," 2 indicates "moderate," 3 indicates "severe," and 4 indicates "very severe." A total score above 3 is generally considered indicative of abnormal swallowing function.
Adverse Events | Within two weeks after surgery, 1 month postoperative, 3 months postoperative, and 6 months postoperative
  At each follow-up visit, adverse events (including adverse drug reactions) were recorded through patient interviews and physical examinations.

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stojadinovic A, Shaha AR, Orlikoff RF, Nissan A, Kornak MF, Singh B, Boyle JO, Shah JP, Brennan MF, Kraus DH. Prospective functional voice assessment in patients undergoing thyroid surgery. Ann Surg. 2002 Dec;236(6):823-32. doi: 10.1097/00000658-200212000-00015. PMID 12454521
- [Result] Xia Y, Zhu Y, Ling L, Xu F, Yang Y, Ye J, Tan W, Chen Z, Liu Q, Wei W, Zhang J, Zhang A, Zhang L, Song E, Gong C. Effect of methylcobalamin on capecitabine induced hand-foot syndrome in patients with HER2 negative early breast cancer: multicentre, double blind, randomised, placebo controlled, phase 3 trial. BMJ. 2025 Sep 11;390:e084290. doi: 10.1136/bmj-2025-084290. PMID 40935571
- [Result] Nishimoto S, Tanaka H, Okamoto M, Okada K, Murase T, Yoshikawa H. Methylcobalamin promotes the differentiation of Schwann cells and remyelination in lysophosphatidylcholine-induced demyelination of the rat sciatic nerve. Front Cell Neurosci. 2015 Aug 4;9:298. doi: 10.3389/fncel.2015.00298. eCollection 2015. PMID 26300733
- [Result] Kim HA, Mindos T, Parkinson DB. Plastic fantastic: Schwann cells and repair of the peripheral nervous system. Stem Cells Transl Med. 2013 Aug;2(8):553-7. doi: 10.5966/sctm.2013-0011. Epub 2013 Jul 1. PMID 23817134
- [Result] Stoll G, Muller HW. Nerve injury, axonal degeneration and neural regeneration: basic insights. Brain Pathol. 1999 Apr;9(2):313-25. doi: 10.1111/j.1750-3639.1999.tb00229.x. PMID 10219748
- [Result] Zhou T, Wang X, Zhang J, Zhou E, Xu C, Shen Y, Zou J, Lu W, Su K, Huang W, Yi H, Yin S. Global burden of thyroid cancer from 1990 to 2021: a systematic analysis from the Global Burden of Disease Study 2021. J Hematol Oncol. 2024 Aug 27;17(1):74. doi: 10.1186/s13045-024-01593-y. PMID 39192360